CLINICAL TRIAL: NCT00591110
Title: Project inCharge: Increasing the Rate of Comprehensive Eye Care Utilization by Older African Americans Through Community-Based Eye Health Education Program
Acronym: inCharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Cynthia Owsley, Nathan E. Miles Chair of Ophthalmology, Vice Chair for Clinical Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X060908004
Record Dates: First submitted 2007-12-21; First posted 2008-01-11 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Eye Disease; Eye Care; Vision
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Educational intervention communicating practical information about vision, eye conditions and eye care.
  Interventions: Behavioral: Eye care education
- 2 (Sham Comparator)
  Interventions: Behavioral: Social-contact control

INTERVENTIONS:
Behavioral: Eye care education — Participants will receive an educational intervention communicating practical information about vision, eye conditions and eye care pertinent to the older African American population
  Arms: 1
Behavioral: Social-contact control — Participants receive an engaging informational session on a non-health related topic
  Arms: 2

SUMMARY:
The study design is a randomized intervention evaluation. Ten senior centers in predominately African American communities in the Birmingham, Alabama will be selected as sites for the educational intervention. Five centers will be randomly assigned to receive an educational intervention communicating practical information about vision, eye conditions and eye care as pertinent to the older African American population. The other five centers will serve as social-contact controls, where participants will receive an engaging information session on a non-health related topic. The primary outcome of interest is the change in percentage of persons receiving comprehensive eye care from pre- to post- intervention. The secondary outcomes are the process outcomes of improvement in knowledge, attitudes, and values about vision, eye conditions, and eye care.

ELIGIBILITY:
Inclusion Criteria:

* African Americans ages >=60 years residing in the communities targeted for intervention or control activities

Exclusion Criteria:

* Persons who do not speak English, persons who are not community-dwelling.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of persons receiving comprehensive eye care from pre- to post- intervention | 6 months

SECONDARY OUTCOMES:
Improvement in knowledge, attitudes, and values about vision, eye conditions, and eye care and reduction in perceived barriers to care. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owsley, PhD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Owsley C, McGwin G Jr, Searcey K, Weston J, Johnson A, Stalvey BT, Liu B, Girkin CA. Effect of an eye health education program on older African Americans' eye care utilization and attitudes about eye care. J Natl Med Assoc. 2013 Spring;105(1):69-76. doi: 10.1016/s0027-9684(15)30087-0. PMID 23862298